CLINICAL TRIAL: NCT01164787
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-sequence, Two-period, Single-dose, Crossover Comparative Bioequivalence Study of Trandolapril 4 mg Tablets of Dr. Reddy's Laboratories Limited and Mavik® 4 mg Tablets of Abbott Laboratories, in Healthy, Adult, Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Trandolapril 4 mg Tablets of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Mr. M.S. Mohan/ Vice President R & D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CL-028-TRAN-2006
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Trandolapril
MeSH Terms: interventions — trandolapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trandolapril (Experimental): Trandolapril 4 mg Tablets of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Trandolapril
- Mavik® (Active Comparator): Mavik® 4 mg Tablets of Abbott Laboratories, USA.
  Interventions: Drug: Mavik

INTERVENTIONS:
Drug: Trandolapril — Trandolapril 4 mg Tablets of Dr. Reddy's Laboratories Limited
  Other Names: Mavik® 4 mg Tablets
  Arms: Trandolapril
Drug: Mavik — Mavik® 4 mg Tablets of Abbott Laboratories, USA.
  Arms: Mavik®

SUMMARY:
The purpose of this study is

* To compare the single oral dose bioavailability of test product, Trandolapril 4 mg Tablets of Dr. Reddy's and Mavik® 4 mg Tablet of Abbott Laboratories, in healthy, adult, human subjects, under fed conditions to assess bioequivalence.
* To monitor adverse events and ensure safety of subjects.

DETAILED DESCRIPTION:
An open label, randomised, two-treatment, two-sequence, two-period, two-way cross-over,single-dose bioequivalence study of Trandolapril4 mg Tablets manufactured by Dr. Reddy's Laboratories Ltd., Generics, India comparing with the Mavik® 4 mg Tablets (containing trandolapril 4 mg) manufactured by Abbott Laboratories, North Chicago, IL 60064, US; in healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human subjects within the age range of 18 to 45 years
* Non-smokers since at least six months
* Willingness to provide written informed consent to participate in the study
* Body-mass index of ≥ 18.5 kg/m2 and ≤24.9 kg/m2, with body weight not less than 50 kg
* Absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluations, medical history or physical examination during the screening Normal 12-lead ECG or one with abnormality considered to be clinically insignificant Normal chest X-ray PA view Comprehension of the nature and purpose of the study and compliance with the requirement of the Protocol
* Female Subjects

  * of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm,intrauterine device (IUD), or abstinence, or
  * postmenopausal for at least 1 year, or
  * surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject

Exclusion Criteria:

* Personal/family history of allergy or hypersensitivity to Trandolapril or allied drugs
* Past history of anaphylaxis or angioedema
* Any major illness in the past three months or any clinically significant ongoing chronic medical illness e.g. congestive heart failure, hepatitis, pancreatitis etc.
* Presence of any clinically significCint abnormal values during screening e.g. significant abnormality of Liver Function Test (LFT), Renal (kidney) Function Test (RFT), etc.
* Any cardiac, renal or liver impairment, any other organ or system impairment
* History of seizure or psychiatric disorders
* Presence of disease markers of HIV 1 and 2, and hepatitis B and C virus
* Consumption of alcohol for more than two years, or consumption of more than three alcoholic drinks per day or consumption of alcohol within 48 hours prior to dosing and during the study [one drink is equal to one unit of alcohol [one glass wine, half pint beer, and one measure (one ounce) of spirit).
* Consumption of xanthine containing derivatives (coffee, tea, cola drinks, chocolate) within 48 hours before check-in of each period
* Use of any recreational drug or a history of drug addiction
* Participation in any clinical trial within the past 3 months
* Inaccessibility of veins in left and right arm
* Donation of blood (one unit or 350 mL) within 3 months prior to receiVing the first dose of study medication
* Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking from 48 hours before dosing and until the completion of the study.
* Receipt of any prescription drug therapy within four weeks or over-the-counter (OTC) drugs within two weeks prior to receiving the first dose of study medication or repeated use of drugs within the last four weeks
* An unusual diet, for whatever reason e.g. low sodium diet, for two weeks prior to receiving any medication and through out subject's participation in the study
* Consumption of grapefruit- containing food or beverages within 10 days prior to receiving the first dose of study medication in both the periods
* Recent history of dehydration from diarrhoea, vomiting or any other reason within a period of 24 hours prior to the study
* Female subjects who are pregnant or who are able (women with child bearing potential) to become pregnant during the study will not be allowed to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2006-03; Primary Completion 2006-04 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Umesh Dhakate, M.B.B.S, Principal Investigator — Wellquest Clinical Research
Locations (1):
- Wellquest Clinical Research, Mumbai, Maharashtra, India